CLINICAL TRIAL: NCT04240587
Title: Intranasal Neurostimulation for the Treatment of Neurosensory Abnormalities in CL Wearers (INTAC)
Acronym: INTAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrollment of study participants
Sponsor: Tufts Medical Center (Other)
Collaborators: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000080
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Contact Allergy; Neuropathic Pain
Keywords: Contact Lens Discomfort
MeSH Terms: conditions — Dermatitis, Allergic Contact; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TrueTear™ intranasal neurostimulator (ITN) Active Arm (Active Comparator): TrueTear™ intranasal neurostimulator (ITN) with active tips - The tips carry the current from the base to the nasociliary nerve.
  Interventions: Device: TrueTear™ intranasal neurostimulator (ITN)
- TrueTear™ intranasal neurostimulator (ITN) Placebo/Sham Arm (Placebo Comparator): TrueTear™ intranasal neurostimulator (ITN) with sham tips - The "sham" tips and do not properly carry the current.
  Interventions: Device: TrueTear™ intranasal neurostimulator (ITN)

INTERVENTIONS:
Device: TrueTear™ intranasal neurostimulator (ITN) — The ITN delivers small electrical currents to the inner cavity of the nose, gently activating nerves that stimulate the body's natural tear production system. Those in the ITN "active" arm will receive the active tips which contain the current from the base to the nasociliary nerve. Those in the ITN "sham" arm will receive tips without the current.

SUMMARY:
To find out if the use of an intranasal tear neurostimulator (ITN), may be useful in decreasing the pain symptoms felt by patients who experience contact lens discomfort.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age at screening visit
* Ocular Surface Disease Index (OSDI) score of less than 12 (without contact lens wear)
* Contact Lens Dry Eye Questionnaire (CLDEQ)-8 score of greater than 12.18
* Regular contact lens wearer who wears them less than 6 hours per day due to discomfort
* The presence of at least one microneuroma on in vivo confocal microscopy
* Self-reported good compliance with healthy contact lens regimen (replace contact lenses per manufacturer's recommendations, use of multipurpose or hydrogen peroxide contact lens solution nightly)
* Have had an eye exam within the last two years that included dispense of a contact lens prescription
* Proparacaine drops relieve at least 75% of ocular symptoms to ensure that patients do not have centralized neuropathic corneal pain
* If a soft lens wearer, use a contact lens that was released within the last 15 years

Exclusion Criteria:

* Use of topical drops other than artificial tear substitutes
* Ocular surgery or other ocular disease within 3 months prior to study enrollment
* Concurrent ocular disease that may impact results
* Have dry eye (as defined by 2 or more of the parameters below)

  * Schirmer's wetting test < 10mm
  * TBUT <7sec
* NEI scale corneal staining of 4 out of 15 at the time of enrollment
* Improper CL fit
* No microneuroma by in vivo confocal microscopy
* Overnight wear within 1 month of screening visit
* Use of colored or cosmetic lenses
* Contra-indication to ITN

  * Chronic or recurrent epistaxis, coagulation disorders.
  * Nasal or sinus surgery or significant trauma to the nose.
  * Cardiac demand pacemaker, implanted defibrillator, or other implanted electronic device in the head or neck.
  * Chronic or recurrent nosebleeds
  * Bleeding disorder
  * Known hypersensitivity (allergy) to the hydrogel material
  * Disabling arthritis, neuropathy, or limited motor coordination affecting self-handling of the device.
  * History of migraines
  * Under 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the decrease in microneuromas by means of in vivo confocal microscopy (IVCM) among CLD subjects following treatment | 3 months
To measure the changes in the level of discomfort/pain after instillation of hyperosmolarity drops among CLD subjects following treatment | 3 months
To measure changes in Contact Lens Dry Eye Questionnaire (CLDEQ)-8 among CLD subjects using ITN. | 3 months

SECONDARY OUTCOMES:
To access the corneal dendritic cells (DC) density by means of IVCM among CLD subjects before and after treatment. | 3 months
To evaluate the change in wearing time and comfortable wearing time from baseline to the final visit. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No